CLINICAL TRIAL: NCT02678026
Title: Pessary as Adjunctive Therapy to Cerclage for the Prevention of Preterm Birth
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no enrollment
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Medical Doctor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111/888
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical Pessary (Experimental): Cervical pessary is a medical device used to treat an incompetent (or insufficient) cervix (cervix starts to shorten and open too early).
  Women will receive pessary soon after UIC
  Interventions: Device: Cervical pessary
- No intervention (No Intervention): No treatment

INTERVENTIONS:
Device: Cervical pessary — Cervical pessary is a medical device used to treat an incompetent (or insufficient) cervix (cervix starts to shorten and open too early). Early in the pregnancy a round silicone pessary is placed at the opening to the cervix to close it, and then remove late in the pregnancy when the risk of a preterm birth has passed.
  Arms: Cervical Pessary

SUMMARY:
Cervical cerclage was devised in the 1950's for women with prior early preterm births (PTB) who developed a dilated cervix detected by manual exam in the second trimester. In contemporary practice, there are three possible indications for cerclage. History-indicated cerclage (HIC) is defined as a cerclage placed usually between 12-15 weeks based solely on poor prior obstetrical history, e.g. multiple second trimester losses due to painless dilatation. Ultrasound-indicated cerclage (UIC) is defined as a cerclage placed usually between 16-23 weeks for transvaginal ultrasound (TVU) cervical length (CL) < 25mm in a woman with a prior spontaneous PTB. Physical-exam indicated is defined as a cerclage placed usually between 16-23 weeks because of cervical dilatation of 1 or more centimeters detected on physical (manual) examination.

Randomized trials and meta-analysis of these have shown that UIC is associated with significant reduction in PTB and improved neonatal outcome, whereas evidence of efficacy for history-indicated cerclage and physical exam-indicated cerclage is limited. In the United States, the national data shows that the rate of cerclage has decreased in the last few years. The indications of placement of cerclage have recently changed, and so it is important to evaluate how many women are getting this procedure. With the recent completion of clinical trials, it is plausible that obstetricians and perinatologists may have become more selective in terms of the best candidates for cerclage.

The aim of this RCT is to evaluate the efficacy of cervical pessary in prevention of PTB as adjuctive therapy in women with UIC

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Singleton gestations
* Women with prior preterm birth and with short cervical length (TVU CL <25 mm) who underwent UIC

Exclusion Criteria:

* multiple gestation
* Ruptured membranes
* Lethal fetal structural anomaly
* Fetal chromosomal abnormality
* Vaginal bleeding
* Suspicion of chorioamnionitis
* Ballooning of membranes outside the cervix into the vagina
* Painful regular uterine contractions
* Labor
* Placenta previa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01-01; Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Preterm delivery | Less than 34 weeks gestation

SECONDARY OUTCOMES:
Gestational age at delivery | Time of delivery
Birth weight | Time of delivery
Spontaneous preterm birth rates | Less than 24, 28, 34 and 37 weeks gestation
Spontaneous rupture of membranes | Less than 34 weeks gestation
Type of delivery: rate of cesaran delivery, vaginal delivery and operative vaginal delivery | Time of delivery
Neonatal death | Between birth and 28 days of age
Composite adverse neonatal outcome | Between birth and 28 days of age
  Includes necrotizing enterocolitis, intraventricular hemorrhage (grade 3 or higher), respiratory distress syndrome, bronchopulmonary dysplasia (BPD), retinopathy, blood-culture proven sepsis and neonatal death
Admission to neonatal intensive care unit | Between birth and 28 days of age
Chorioamnionitis | Time of delivery
significant adverse maternal effects | Time of delivery
  Includes heavy bleeding, injury (eg erosion; fistula; etc) to vagina; injury (eg erosion; fistula; etc) to bladder, cervical tear and uterine rupture
Intolerance to pessary | prior to delivery
  Defined as request for removal secondary to discomfort and/or discharge
Preterm delivery | Less than 24, 28 and 37 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

REFERENCES:
- [Derived] Eleje GU, Eke AC, Ikechebelu JI, Ezebialu IU, Okam PC, Ilika CP. Cervical stitch (cerclage) in combination with other treatments for preventing spontaneous preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2020 Sep 24;9(9):CD012871. doi: 10.1002/14651858.CD012871.pub2. PMID 32970845